CLINICAL TRIAL: NCT07151625
Title: To Complement or Not Complement- Is Protein Complementation at Each Meal Necessary When Consuming Plant-based Diets?
Brief Title: Protein Complementation of Plant-based Diets.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Glenda Courtney-Martin, Senior Associate Scientist- Translational Medicine, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 3667; PJT-198014 (Other Grant/Funding Number: CANADIAN INSTITUTE FOR HEALTH RESEARCH)
Record Dates: First submitted 2025-08-18; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Each Participant Will be Studied Over 5 Dietary Periods, Each Over 9d
Keywords: protein complementation; whole body protein turnover; protein synthesis; protein breakdown; protein balance; humans
MeSH Terms: interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- protein synthesis, breakdown and balance assessed after exposure to 5 diets consumed over 9d (Other)
  Interventions: Other: Diet, whole food provided to participants over 5 x 9 day period; Other: Diet

INTERVENTIONS:
Other: Diet, whole food provided to participants over 5 x 9 day period — 5 diets provided to participants over 9 days each and whole body protein synthesis, protein breakdown and protein balance assessed after each period.
Other: Diet — 5 different diet types

SUMMARY:
Amino acids are the building blocks of proteins which are needed by the body for growth, and bodily functions. If even one amino acid is in short supply, this will negatively affect growth and various functions in the body. Animal foods like meat, fish and chicken contain all the amino acids needed by the body in the correct proportion. These foods are considered high quality protein foods. However plant proteins like lentils, wheat, rice are low in at least one amino acid. This means that plant proteins are considered low quality proteins.

Data from the investigators lab and others show that when eating plant foods, combining grains and legumes like rice and beans, peanut butter and bread, (protein complementation) will provide a complete protein which contains all the amino acids needed by the body. However, some maintain that it is not necessary to combine foods like grains and legumes in the same meal as long as all the amino acids are consumed within a 24h period. This has never been tested.

The goal of this study is to compare the effects non-complementation to protein complementization on whole body protein metabolism in young and older adults.

DETAILED DESCRIPTION:
Complementation of plant proteins with complementary amino acid profile (cereal grain + legume) in each meal can improve the protein quality of plant based diets. However, some maintain that if a variety of plant foods are consumed throughout the day, all essential amino acids are provided and protein complementation at each meal is unnecessary. This assumption has NEVER been tested, yet it forms the basis of current expert recommendations for vegetarian diets. Evidence from the investigators lab and others demonstrate that there is no storage pool of amino acids in the body; when one amino acid is deficient in the diet for protein synthesis, all others are in relative excess and are oxidized resulting in poor growth and lower rates of protein synthesis. Therefore, current recommendations for plant based diet consumption could be misleading.

Skeletal muscle plays an important role in the adaptations of body proteins to nutritional changes and during stress. Therefore, knowledge of skeletal muscle response to changes in dietary protein intake from animal to plant based protein is an important prerequisite to understand the body's capacity, especially in the elderly, to adapt to alterations in dietary protein quality from animal to plant based, whether in complementation or non-complementation fashion. The contribution of skeletal muscle to protein breakdown is calculated by measuring urinary 3-methylhistidine. This amino acid is produced in muscle from post-translational modification of histidine and released from actin and myosin. It is not reutilized for protein synthesis but is excreted in the urine. Therefore, the urinary output of 3-methylhistidine is a quantitative index of daily muscle protein breakdown.

Objectives:

1. To assess whole-body protein metabolism (WBPM) (protein synthesis, protein breakdown and protein balance) using a single dose [15N]glycine and measuring cumulative excretion of [15N]urea in urine in human adult consuming a PB diet provided in a complementary or non-complementary fashion in males and females 18 -39, 60-69 and 70-79 years and
2. To assess the contribution of skeletal muscle to protein breakdown by measuring urinary 3-methyhistidine.

Hypothesis:

Protein synthesis and balance will be lower, but breakdown will be higher in the non-complementation PB diets compared to omnivorous diet (control) and lacto-vegetarian diet.

ELIGIBILITY:
Inclusion Criteria:

* 1) Young Adults:
* Adults, age 18 - 39 yrs, Healthy with no known clinical condition which would affect protein or AA metabolism, ex. Diabetes, Stable Body Weight (no more than 5 lb weight loss or gain in the past 3 months)
* Not on any medications that could affect protein or amino acid metabolism e.g. steroids.
* Fasting blood glucose, hemoglobin A1C (HbA1c), urea and creatinine within normal ranges for age.

  2) Older Adults:
* Adults, aged 60-69 and 70-79 years, Healthy with no known clinical condition which would affect protein or AA metabolism, ex. Diabetes, Stable Body Weight (no more than 5 lb weight loss or gain in the past 3 months)
* Not on any medications that could affect protein or amino acid metabolism e.g. steroids,
* Fasting blood glucose, hemoglobin A1C (HbA1c), urea and creatinine within normal ranges for age.

Exclusion Criteria:

* Unwillingness to participate or unable to tolerate the diet
* Recent history of weight loss within the last 3 months or on a weight reducing diet Inability to tolerate study diets (ex. Allergy to ingredients).
* Significant caffeine consumption (>2 cups per day)
* Significant alcohol consumption (>1 drink per day i.e. 1 beer or ½ glass of wine).
* Fasting blood glucose, hemoglobin A1C (HbA1c), urea and creatinine outside of normal ranges for age.
* On medications known to affect protein and AA metabolism, renal failure, liver disease, unable to ambulate independently.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Whole-body protein metabolism (WBPM): protein synthesis, protein breakdown and protein balance. | 9 days
  Protein synthesis, protein breakdown and protein balance (synthesis-breakdown) will be calculated from urinary urea enrichments using standard equations previously used by the investigators and others. The skeletal muscle content of 3-methylhistidine will be used to compute the rate of whole body muscle protein breakdown from the daily urinary excretion of the 3-methylhistidine. Non-muscle component will be computed by subtracting the muscle protein breakdown (3-methylhistidine) from the whole-body protein breakdown obtained from the urine [15N]urea data.

CONTACTS AND LOCATIONS:
Overall Officials: Glenda Courtney-Martin, PhD, RD, Principal Investigator — Research Institute, The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers unless doing a metanalysis and data is requested. The information will be uploaded as per the ICMJE requirements at the end of the study.